CLINICAL TRIAL: NCT01251965
Title: A Phase I/II Study to Determine the Safety and Efficacy of Ruxolitinib, a JAK1/JAK2 Inhibitor, in Subjects With Relapsed or Refractory Acute Leukemia
Brief Title: Phase l/II Study of Ruxolitinib for Acute Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped by the principal investigator due to nonsatisfactory clinical benefit even in patients treated at the highest dose (200 mg ).
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0450; NCI-2011-02439 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Leukemia
Keywords: Relapsed Acute Leukemia; Acute myeloid leukemia; AML; Acute lymphocytic leukemia; ALL; Ruxolitinib; Jakafi; INC424; INCB018424
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Phase I is a standard 3+3 design and will be used to determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD), and no formal evaluation of efficacy (response rate will be implemented. Patients in Phase I part who were treated at the MTD will be included toward patients assessed for response in the phase II stage.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ruxolitinib 50 mg BID (Experimental): Phase I - Starting dose of Ruxolitinib 50 mg by mouth twice a day for 28 day cycle.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib 100 mg BID (Experimental): Phase I dose of Ruxolitinib 100 mg by mouth twice a day for 28 day cycle.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib 200 mg BID (Experimental): Phase I dose of Ruxolitinib 200 mg by mouth twice a day for 28 day cycle.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Phase I - Starting dose of 50 mg by mouth twice a day for 28 day cycle.
  Phase II - MTD reached in Phase I.
  Other Names: Jakafi; INCBO18424; INC424

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of ruxolitinib that can be given to patients with acute leukemia and to learn if the study drug can help control the disease. The safety of the drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Ruxolitinib is designed to block a gene mutation that may be important in cancer cell growth and survival. By blocking the gene mutation, this may cause the cancer cells to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 30 participants will be enrolled in the Phase I portion of the study, and up to 136 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of ruxolitinib you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of ruxolitinib. Each new group will receive a higher dose of ruxolitinib than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of ruxolitinib is found.

If you are enrolled in the Phase II portion, you will receive ruxolitinib at the highest dose that was tolerated in the Phase I portion or at a lower dose.

Study Drug Administration:

You will take ruxolitinib tablet(s) by mouth 2 times a day on Days 1-28 of each 28-day study cycle.

You will be asked to keep a diary to record the doses taken. You will be asked to bring your diary and any unused drug to your next visit.

Study Visits:

On Days 1, 7, 14, and 21 of Cycle 1:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked about any treatments you may have had, any other drugs you may be taking, and any side effects you may be having.
* On Day 14 only, you will have a bone marrow aspiration performed to check the status of the disease.

On Day 1 of Cycle 2:

* You will have a physical exam.
* You will be asked about any treatments you may have had, any other drugs you may be taking, and any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have a bone marrow aspiration performed to check the status of the disease.

During Cycles 2 and beyond, blood (about 2 teaspoons) will be drawn for routine tests at least every 1-2 weeks. This blood may be drawn at a clinic close to your home.

On Day 1 of Cycles 3, 6, 9, and beyond:

* You will have a physical exam.
* You will be asked about any treatments you may have had, any other drugs you may be taking, and any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have a bone marrow aspiration performed to check the status of the disease. On Day 1 of Cycle 3, this will only be done if your doctor thinks it is needed.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over once you have completed the end-of-study visit and the follow-up call.

End-of-Study Visit:

After your last dose of study drug, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* You will be asked about any treatments you may have had, any other drugs you may be taking, and any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have a bone marrow aspiration performed to check the status of the disease.

Follow-Up:

About one month after your end-of-study visit, the study staff will call and ask about any side effects you may be having. This call should last about 5 minutes.

This is an investigational study. Ruxolitinib is FDA approved and commercially available for the treatment of intermediate or high-risk myelofibrosis, including primary myelofibrosis, post-polycythemia vera (post-PV) myelofibrosis and post-essential thrombocythemia (post-ET) myelofibrosis. Its use to treat acute leukemia is investigational.

Up to 166 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Must be >14 years of age
2. Must be diagnosed with refractory or relapsed AML or ALL.
3. Must have adequate organ function as demonstrated by the following: o Alanine Aminotransferase (ALT) (SGOT) and/or Aspartate Aminotransferase (AST) (SGPT) equal to or less than 1.5x upper limit of normal o Serum creatinine equal to or less than 2.5 mg/dL
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
5. At least 2 weeks from prior leukemia-directed treatment to starting treatment drug (except for hydroxyurea, which is allowed if clinically indicated but should be stopped after 2 weeks of receiving study drug, and glucocorticoids, which are allowed but should be stopped upon starting treatment drug).
6. Treatment-related toxicities from prior therapies must have resolved to Grade equal to or less than 1 (except for peripheral neuropathy, which should resolve to grade equal to or less than 2)
7. No active malignancies with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
8. Females of childbearing potential (FCBP)(A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) must have negative pregnancy test. FCBP and males participating in the study must agree to use a reliable form of contraception or to practice complete abstinence from heterosexual intercourse while participating in the study and for at least 28 days after discontinuation from the study. If pregnancy or a positive pregnancy test does occur in a study subject, treatment with the study drug must be immediately discontinued.

Exclusion Criteria:

1. Known positive status for HIV, or known active hepatitis A, B, or C infection.
2. Any serious medical condition or psychiatric illness that would prevent, (as judged by the treating physician) the subject from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
3. Pregnant or lactating females.
4. Acute promyelocytic leukemia
5. Concurrent use of strong inducers or strong inhibitors of cytochrome P450 3A4 (CYP3A4). Strong inducers are rifampin and St. John's Worth. Strong inhibitors are HIV-antivirals, clarythromycin, itraconazole, ketoconazole, nefazodone, and telithromycin.
6. Participating in any other research trial.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Pemmaraju N, Kantarjian H, Kadia T, Cortes J, Borthakur G, Newberry K, Garcia-Manero G, Ravandi F, Jabbour E, Dellasala S, Pierce S, Verstovsek S. A phase I/II study of the Janus kinase (JAK)1 and 2 inhibitor ruxolitinib in patients with relapsed or refractory acute myeloid leukemia. Clin Lymphoma Myeloma Leuk. 2015 Mar;15(3):171-6. doi: 10.1016/j.clml.2014.08.003. Epub 2014 Sep 17. PMID 25441108
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 9, 2010 to September 26, 2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Ruxolitinib 50 mg BID: Phase I starting dose of Ruxolitinib 50 mg by mouth twice a day (BID) for 28 day cycle.
Period: Overall Study
Arm/Group | Ruxolitinib 50 mg BID | Ruxolitinib 100 mg BID | Ruxolitinib 200 mg BID
Started | 4 | 5 | 18
Completed | 3 | 3 | 7
Not Completed | 1 | 2 | 11
Not completed — Participant/physician decision | 1 | 2 | 0
Not completed — Death | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib 50 mg BID | Ruxolitinib 100 mg BID | Ruxolitinib 200 mg BID | Total
Number analyzed (Participants) | 4 | 5 | 18 | 27
Age, Continuous [Median (Full Range); unit: years] | 66 [51 to 69] | 70 [41 to 85] | 71 [55 to 83] | 69 [41 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 9 | 13
  Male | 1 | 4 | 9 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 18 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: MTD defined as highest dose level at which no more than one out of six subject experiences dose limiting toxicity (DLT) during first cycle (28 days) of therapy. A non-hematologic DLT defined as a clinically significant grade 3 or 4 adverse event or abnormal laboratory value (according to Common Toxicity Criteria for Adverse Effects (CTCAE) criteria) assessed as related to study drug (and unrelated to disease progression, intercurrent illness, or concomitant medications) occurring during first 28 days on study. Participants who received at least 80% of the originally assigned doses in the first cycle were evaluable for DLT assessment of each cohort.
Time Frame: End of first 28 day cycle for toxicity
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 50 mg BID | Ruxolitinib 100 mg BID | Ruxolitinib 200 mg BID
Number analyzed (Participants) | 3 | 3 | 7
Participants | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Ruxolitinib
Description: The MTD is defined as the highest dose level at which no more than one out of six subject experiences DLT during the first cycle (28 days) of therapy.
Time Frame: End of first 28 day cycle
Measure: Number; unit: mg
Groups:
- Ruxolitinib: Phase I - Starting dose of Ruxolitinib 50 mg by mouth twice a day for 28 day cycle.
  Phase II - MTD reached in Phase I.
  Ruxolitinib: Phase I - Starting dose of 50 mg by mouth twice a day for 28 day cycle.
  Phase II - MTD reached in Phase I.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 13
mg | NA — The Maximum tolerated dose (MTD) was not determined as there were no dose limiting toxicities (DLT's) observed at the doses tested.

3. Secondary Outcome: Participants With a Response
Description: Response is defined as complete remission (CR) + complete remission with incomplete blood count (CRi) + Hematologic improvement (HI). Response was to be assessed for participants who were evaluated for the Phase II portion of this study. CR is absolute neutrophil count (ANC) >/= 1x109/L and platelet count >/= 100x109/L, absence of leukemia blast cells, normal marrow differential, and complete resolution of extramedullary disease. CRi is CR but platelets are < 100x109/L or ANC is <1x109/L. HI is described by the number of individual, positively affected cell lines without the use of growth factors and/or transfusions (lasting at least 4 weeks).
Time Frame: Up to 1 year
Population: The study was stopped because of a lack of satisfactory clinical benefit, and did not go on to the Phase II portion. Therefore, data were not collected for this outcome measure.
Arm/Group | Ruxolitinib 50 mg BID | Ruxolitinib 100 mg BID | Ruxolitinib 200 mg BID
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected during 28 day cycle, up to 9 cycles.
Arm/Group | Ruxolitinib 50 mg BID | Ruxolitinib 100 mg BID | Ruxolitinib 200 mg BID
Serious Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 18/18
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib 50 mg BID (N=4) | Ruxolitinib 100 mg BID (N=5) | Ruxolitinib 200 mg BID (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cerebral edema and mass (Nervous system disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Fever (General disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Neutropenia (Investigations) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib 50 mg BID (N=4) | Ruxolitinib 100 mg BID (N=5) | Ruxolitinib 200 mg BID (N=18)
Hemoglobin Increased (Investigations) | 1 | 1 | 0
Neutrophils count decreased (Investigations) | 2 | 2 | 6
Platelets decreased (Investigations) | 2 | 3 | 6
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Constiptation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Mucositis (Gastrointestinal disorders) | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Edema: head and neck (General disorders) | 1 | 0 | 2
Edema: limb (General disorders) | 0 | 0 | 1
Alkaline phosphatase Increased (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (ALT) (Investigations) | 1 | 2 | 4
Aspartate aminotransferase increased (AST) (Investigations) | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 2 | 1
Creatinine Increased (Investigations) | 1 | 2 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Central Nervous System Ischemia (Nervous system disorders) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1
Neurology-Other Issues (Nervous system disorders) | 0 | 0 | 1
Speech impairment (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hot Flash (Reproductive system and breast disorders) | 0 | 0 | 1
Infections (Infections and infestations) | 4 | 2 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes